CLINICAL TRIAL: NCT06248723
Title: ItaliaN Study With Tailored Multidomain Interventions to Prevent Functional and Cognitive Decline in Community-dwelling Older Adults
Acronym: IN TeMPO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milano Bicocca (Other)
Collaborators: European Union (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IN TeMPO
Record Dates: First submitted 2023-12-27; First posted 2024-02-08 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Age-related Cognitive Decline
Keywords: Cognitive decline; Dementia; Aging
MeSH Terms: conditions — Cognitive Dysfunction; Dementia | interventions — Exercise; Cognitive Training; Oral Hygiene; Metabolic Networks and Pathways

STUDY DESIGN:
Intervention Model Description: The patients are randomized 1:1 into "active intervention" and "self-guided intervention" parallel groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active intervention arm (Experimental): * Physical exercise regime
  * Mediterranean diet-based nutritional plan
  * Cognitive training
  * Regular medical check-ups
  * Oral hygiene treatments and counseling
  * Counseling on sleep hygiene and treatment
  * Control of cardiovascular, metabolic, and infectious risk factors
  * Adjustment of drug therapy
  * Suggestions for improving social interactions
  Physical exercise and cognitive training interventions will be monitored and partially administered through wearable devices and digital tools. Sleep quality will be monitored through wearable devices. Social interactions will be encouraged through a validated app.
  Interventions: Other: Nutritional intervention; Other: Physical exercise; Other: Cognitive training; Other: Oral hygiene; Other: Sleep quality; Other: Control of cardiovascular, metabolic, and infectious risk factors; Other: Pharmacological evaluation; Behavioral: Socializing
- Self-administered intervention arm (Active Comparator): Subjects in the control group will receive regular health advice in the same domains as the intervention group, via dedicated app and/or access to the dedicated portal on the Age-It website.
  In addition, participants randomized to the self-guided intervention will receive an initial 30-60 minute counseling session on all domains covered by the study, in which guidelines for healthy diet, physical and cognitive activity, benefits of social activity, information on cardiovascular risk factors, as well as sleep, oral hygiene will be explained.
  Subjects will therefore be treated as per normal clinical practice, albeit with the help of dedicated apps and counseling session.
  Interventions: Other: Self-administered interventions

INTERVENTIONS:
Other: Nutritional intervention — The objectives of the dietary intervention will be in accordance with the principles of the Mediterranean diet. Weekly menus will be provided that ensure a balanced intake of the various nutrients, according to the objectives outlined in the study protocol, including a reduction in saturated fatty acids (with proportionately more mono- and polyunsaturated fatty acids), promotion of fiber sources and reduction of sugars, adequate protein and micronutrient intake. They will be accompanied by specific dietary patterns that can be individualized based on weight, comorbidities and personal preferences.
  The need for weight loss or gain will be assessed on an individual basis. Dietary interventions will include group and individual sessions, and will be conducted by dietitians and nutritionists in a harmonized manner among the centers. The first meeting will be in-person and will be held at the subject's clinical center of enrollment. Follow-up will be conducted through online meetings.
  Arms: Active intervention arm
Other: Physical exercise — The physical activity protocol will be geared to the principles of progressive and individualized loading, in group sessions supervised by a physical therapist within gyms for the strength and balance training portion, and in moderate to intense aerobic activities based on individual preferences and characteristics. The physiotherapist will conduct an individual assessment and develop personalized programs for all participants. Exercise sessions will be held 2-3 times a week.
  Arms: Active intervention arm
Other: Cognitive training — Participants will be evaluated through a Cognitive and Psychological Assessment, which will allow measurement of each participant's cognitive functioning and well-being. Computerized cognitive training (CCT) using Brain HeadQuarter (BrainHQ) or similar software will be used as a cognitive intervention. The CCT includes game-based adaptive exercises that target attention, intelligence, memory, navigation, processing speed and social skills. The training will consist of 72 sessions for 24 weeks (about six months), at least three times a week.
  Arms: Active intervention arm
Other: Oral hygiene — Participants will be referred for evaluation at dental hygiene offices. As part of the study, participants will also undergo anticholinergic burden calculation, screening for risk factors for oral diseases (smoking, alcohol), and reduction in the frequency of sugar intake through dietary intervention will be sought.
  Participants will also undergo the Oral Health Assessment Tool rating scale.
  Arms: Active intervention arm
Other: Sleep quality — During the visits, participants' sleep will be assessed, either by clinical interview or by scales. Participants will also have the opportunity to assess their own sleep via wearable devices.
  If sleep hygiene issues are detected, advice based on currently available scientific evidence will be provided. If, on the other hand, a suspicion of sleep disorders, including, for example, obstructive sleep apnea syndrome, restless legs syndrome, insomnia, or Rapid Eye Movement (REM) sleep disorder, is raised from the medical history, participants will be referred to the relevant specialists for diagnosis and treatment of such problems.
  Arms: Active intervention arm
Other: Control of cardiovascular, metabolic, and infectious risk factors — Measurements of blood pressure, weight, BMI, abdominal circumference, and advice on health promotion and healthy lifestyle will be provided. Recommendations on adherence to the Piano Nazionale di Prevenzione Vaccinale (PNPV) will also be provided.
  Arms: Active intervention arm
Other: Pharmacological evaluation — Evaluation of prescriptive appropriateness (STOP&START and Beers criteria) and calculation of anticholinergic burden (ACB calculator) will be carried out by a geriatrician, with rationalization of therapy and, where possible, de-prescribing.
  Arms: Active intervention arm
Behavioral: Socializing — To encourage socialization, proposed activities will be carried out as much as possible in groups of 10-12 people, and outdoor group activities will be suggested on a biweekly basis (e.g., walks in parks). On a monthly basis, the nurse and psychologist will organize motivational and check-up meetings (in recreation centers/via telematics) in order to promote adherence to the protocol, collect questions and stimulate participants.
  Social activity will also be implemented in the context of all interventions, for example through:
  * Physical activity in groups or pairs, including dance or choir activities where possible
  * Opportunities for further cognitive stimulation in groups through games (e.g., chess, cards, etc.)
  * Proposal to cook, eat or shop together
  * Group sessions with dietitian
  Arms: Active intervention arm
Other: Self-administered interventions — Subjects in the control group will receive regular health advice in the same domains as the intervention group, via dedicated app and/or access to the dedicated portal on the Age-It website. Such advice and information will be timed to encourage adherence. In addition, participants randomized to the self-guided intervention will receive an initial counseling session of 30-60 minutes on all domains covered by the study, where guidelines for healthy diet, physical and cognitive activity, benefits of social activity, information on cardiovascular risk factors, as well as sleep, oral hygiene will be explained.
  Subjects will therefore be treated as per normal clinical practice, albeit with the help of dedicated apps and counseling session.
  Arms: Self-administered intervention arm

SUMMARY:
The goal of this interventional non-pharmacological study is to investigate the effects of a multi-domain intervention ( "active intervention"), compared to that followed by normal clinical practice ("self-guided intervention"), in older adults. The primary objective is whether these interventions can prevent functional and cognitive decline in at-risk subjects.

The multi-domain interventions will include physical exercise, a Mediterranean diet-based nutritional plan, cognitive training, regular medical check-ups, oral hygiene treatments and counseling, monitoring and counseling on visual and auditory abilities, counseling on sleep hygiene and treatment, control of cardiovascular, metabolic, and infectious risk factors, adjustment of drug therapy, suggestions for improving social interactions.

DETAILED DESCRIPTION:
The study is multicentric and will include 10 centers. Patients will be enrolled either through their General Practitioners (GPs), which will then refer back to their reference centers, or through the centers themselves.

Patients will undergo a screening visit, which will include a multi-faceted evaluation of cognitive function, physical and functional efficiency, and cardiovascular and cognitive decline risk factors. Procedures to be carried out during the screening visit include:

* Collection of socio-demographic data (age, sex, marital status, cohabitation, level of education, social interactions), clinical details (medical and medication history), and evaluation of inclusion/exclusion criteria
* Assessment of the degree of frailty through the Primary Care Frailty Index (PC-FI)
* Assessment of the presence of increased risk of developing dementia through the Cardiovascular Risk Factors, Aging, and Incidence of Dementia (CAIDE) score
* Assessment of cognitive performance through the General Practitioner assessment of COGnition (GPCOG)
* Assessment of cognitive performance through the Rey Auditory Verbal Learning Test - immediate
* Assessment of functional status by Short Physical Performance Battery (SPPB) tests
* Nonverbal interference tests
* Assessment of cognitive performance through the Rey Auditory Verbal Learning online version (RAVL-T delayed)
* Collection of self-administered scales for cognitive performance assessment through the Test Your Memory - Italian (TYM-I) scale.

Then, eligible patients will be enrolled for the second, active intervention phase of the study, which will include a baseline visit and 3 follow-up visits, at 6, 12, and 18 months.

During these visits, primary and secondary endpoint outcomes will be collected according to protocol.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 or older
* Mild/moderate vulnerability (Primary Care Frailty Index score between 0.07 and 0.21)
* Cardiovascular risk factors, Ageing and Incidence of Dementia (CAIDE) > 6
* Clinical Dementia Rating (CDR) ≤ 0.5
* Presence of increased risk of developing dementia by family history (≥ 1 family member with dementia) and/or at least one modifiable risk factor, with Lifestyle Index ≥2. Lifestyle index evaluation: each "Yes" answer to the following questions = 1 point.

  1. Physical activity less than 2.5 hours per week (defined as physical activity intense enough to lead to sweating and breathlessness)*
  2. Diet: less than 5 servings of fruits and vegetables per day*
  3. Diet: less than 2 servings of fish per week*
  4. Hypertension: diagnosed by a physician or on medication, or Systolic Blood Pressure (SBP)>140 mmHg, or Diastolic Blood Pressure (DBP)>90 mmHg)
  5. Diabetes: type 1 or type 2 diagnosed by a physician, or on medication, or HbA1C ≥7 % in the previous 6 months
  6. Sleep disturbances, depressive symptoms, or mental/physical stress symptoms, for at least 1 month, judged by the physician to be disabling in daily life
  7. BMI ≥ 25 kg/m^2*
  8. Alcohol: > 21 alcohol units/week*. *Based on international and WHO guidelines.
* Informed consent freely given and acquired before the start of the study

Exclusion Criteria:

* Diagnosis of dementia or suspected dementia following the screening visit
* CDR > 0.5
* Residents in residential facilities for the elderly
* Inability to consent to informed consent and/or actively participate in study interventions, according to clinical judgment
* Any condition that prevents safe involvement in the intervention and/or cooperation in the study. For example, a significant neurological or psychiatric condition, including but not limited to brain tumors (benign or malignant), major psychiatric disorders (e.g. current major depressive disorder, schizophrenia, schizoaffective disorder or bipolar disorder), recent brain hemorrhage (parenchymal or subdural), history of concussive head trauma with persistent or significant neurological outcomes, known morpho-structural abnormalities in the brain, active alcohol/drug abuse, active uncontrolled disease of any major organ system; history within the last six months of any acute disease of a major organ system requiring emergency care or hospitalization, including revascularization procedures; severe renal or hepatic insufficiency; unstable or poorly controlled diabetes mellitus, hypertension, or heart failure; malignant neoplasms within the past 3 years (except basal cell carcinoma or squamous cell carcinoma in situ of the skin or localized prostate adenocarcinoma in male participants); any clinically relevant abnormality in blood parameters; severe loss of vision, smar or communication ability, such as to prevent cooperation.
* Enrollment in other trials
* High performance on screening memory tests: RAVL-T immediate score >48 (score ranges 0-75), RAVL-T delayed >10 (score ranges 0-15)
* Planned transfers from the municipality of residence during the duration of the study for a duration longer than 2 weeks.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1340 (Estimated)
Dates: Start 2024-07-16 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Modified Neuropsychological Test Battery (mNTB) score | The score will be taken at Baseline visit (Day 0 of second phase, which should be indicatively within 30 days of Screening visit), at Month 6 follow up, Month 12 follow up, and Month 18 follow up. The tests take around 90 minutes overall.
  Participants will be scored through the mNTB to assess their cognitive state at baseline and cognitive changes at follow-ups. The mNTB score is a composite score for a battery of 14 tests total. The outcome measure is a z-score, it has no minimum or maximum value. A higher score means a better outcome.

SECONDARY OUTCOMES:
Short Physical Performance Battery (SPPB) score | The score will be taken at Day 0 Screening visit, at Baseline visit (Day 0 of second phase, which should be indicatively within 30 days of Screening visit), at Month 6, Month 12, and Month 18 follow-ups.
  Minimum score: 0, maximum score: 12, a higher score means a better performance.
4-m gait speed test - time | The test will be repeated at Baseline visit (Day 0 of second phase, which should be indicatively within 30 days of Screening visit), at Month 6, Month 12, and Month 18 follow-ups.
  Time needed to walk 4 meters (in seconds). A higher time means a worse performance.
4-m gait speed test - speed | The test will be repeated at Baseline visit (Day 0 of second phase, which should be indicatively within 30 days of Screening visit), at Month 6, Month 12, and Month 18 follow-ups.
  Walking speed (in meters per second). A higher speed means a better performance.
Hand grip test | The test will be repeated at Baseline visit (Day 0 of second phase, which should be indicatively within 30 days of Screening visit), at Month 6, Month 12, and Month 18 follow-ups.
  Hand grip strength measured (in kilograms) with a hand dynamometer. A higher result means a better performance.
Activities of Daily Living (ADL) index score | The score will be taken at Day 0 Screening visit, at Baseline visit (Day 0 of second phase, which should be indicatively within 30 days of Screening visit), at Month 6, Month 12, and Month 18 follow-ups..
  Minimum score: 0, maximum score: 6, a higher score means a better performance.
Instrumental Activities of Daily Living (IADL) scale score | The score will be taken at Day 0 Screening visit, at Baseline visit (Day 0 of second phase, which should be indicatively within 30 days of Screening visit), at Month 6, Month 12, and Month 18 follow-ups.
  Minimum score: 0, maximum score: 8, a higher score means a better performance.
Barthel Index score | The score will be taken at Baseline visit (Day 0 of second phase, which should be indicatively within 30 days of Screening visit), at Month 6, Month 12, and Month 18 follow-ups.
  Minimum score: 0, maximum score: 100, a higher score means a better performance.
14-item Resilience Scale (RS-14) score | The score will be taken at baseline, at Month 6, Month 12, and Month 18 follow-ups.
  Minimum score: 14, maximum score: 98, a higher score means a better outcome.
Number of falls taken | Through study completion, an average of 2 years.
  A higher number of falls means a worse outcome.
Number of hospital admissions | Through study completion, an average of 2 years.
  A higher number of hospital admissions means a worse outcome.
Number of visits to general practitioner | Through study completion, an average of 2 years.
  The number does not indicate a better or worse outcome. It is only informative.
Geriatric Depression Scale (GDS) score | The score will be taken at Baseline visit (Day 0 of second phase, which should be indicatively within 30 days of Screening visit), at Month 6, Month 12, and Month 18 follow-ups.
  Minimum: 0, maximum: 15, a higher score indicates a worse outcome.
UCLA Loneliness Scale (UCLA-LS) score | The score will be taken at Baseline visit (Day 0 of second phase, which should be indicatively within 30 days of Screening visit), at Month 6, Month 12, and Month 18 follow-ups.
  Minimum: 20, maximum: 80, a higher score indicates a worse outcome.
Psychological General Well Being Index (PGWBI) score | The score will be taken at Baseline visit (Day 0 of second phase, which should be indicatively within 30 days of Screening visit), at Month 6, Month 12, and Month 18 follow-ups.
  Minimum: 0, maximum: 110, a higher score indicates a worse outcome.
World Health Organization Quality Of Life Questionnaire - Brief (WHO-QOL-Brief) score - Physical Health | The score will be taken at Baseline visit (Day 0 of second phase, which should be indicatively within 30 days of Screening visit), at Month 6, Month 12, and Month 18 follow-ups.
  Minimum: 0, maximum: 100, a higher score means a better outcome.
World Health Organization Quality Of Life Questionnaire - Brief (WHO-QOL-Brief) score - Psychological Health | The score will be taken at Baseline visit (Day 0 of second phase, which should be indicatively within 30 days of Screening visit), at Month 6, Month 12, and Month 18 follow-ups.
  Minimum: 0, maximum: 100, a higher score means a better outcome.
World Health Organization Quality Of Life Questionnaire - Brief (WHO-QOL-Brief) score - Social Relationships | The score will be taken at Baseline visit (Day 0 of second phase, which should be indicatively within 30 days of Screening visit), at Month 6, Month 12, and Month 18 follow-ups.
  Minimum: 0, maximum: 100, a higher score means a better outcome.
World Health Organization Quality Of Life Questionnaire - Brief (WHO-QOL-Brief) score - Environment | The score will be taken at Baseline visit (Day 0 of second phase, which should be indicatively within 30 days of Screening visit), at Month 6, Month 12, and Month 18 follow-ups.
  Minimum: 0, maximum: 100, a higher score means a better outcome.
World Health Organization Quality Of Life Questionnaire - Brief (WHO-QOL-Brief) score - Quality of Life | The score will be taken at Baseline visit (Day 0 of second phase, which should be indicatively within 30 days of Screening visit), at Month 6, Month 12, and Month 18 follow-ups.
  Minimum: 1, maximum: 5, a higher score means a better outcome.
World Health Organization Quality Of Life Questionnaire - Brief (WHO-QOL-Brief) score - Health Satisfaction | The score will be taken at Baseline visit (Day 0 of second phase, which should be indicatively within 30 days of Screening visit), at Month 6, Month 12, and Month 18 follow-ups.
  Minimum: 1, maximum: 5, a higher score means a better outcome.
Pittsburgh Sleep Quality Index (PSQI) score | The score will be taken at Baseline visit (Day 0 of second phase, which should be indicatively within 30 days of Screening visit), at Month 6, Month 12, and Month 18 follow-ups.
  Minimum: 0, maximum: 21, a higher score means a worse outcome.
Mini Nutritional Assessment-Short Form (MNA-SF) score | The score will be taken at Baseline visit (Day 0 of second phase, which should be indicatively within 30 days of Screening visit), at Month 6, Month 12, and Month 18 follow-ups.
  Minimum: 0, maximum: 14, a higher score means a better outcome.
Mediterranean Diet Scale (MDScale) score | The score will be taken at Baseline visit (Day 0 of second phase, which should be indicatively within 30 days of Screening visit), at Month 6, Month 12, and Month 18 follow-ups.
  Minimum: 0, maximum: 9, a higher score means a better outcome.
Framingham Risk Score | The score will be taken at Baseline visit (Day 0 of second phase, which should be indicatively within 30 days of Screening visit), at Month 6, Month 12, and Month 18 follow-ups.
  Measured in percentage %, 0-100%. A higher percentage indicates a higher cardiovascular risk (worse outcome).
Cognitive Reserve Index questionnaire (CRIq) score | The score will be taken at Baseline visit (Day 0 of second phase, which should be indicatively within 30 days of Screening visit), at Month 6, Month 12, and Month 18 follow-ups.
  z-score without a maximum or minimum value, a higher z-score means a better outcome.
Intrinsic Motivation Inventory (IMI) score | The score will be taken at Baseline visit (Day 0 of second phase, which should be indicatively within 30 days of Screening visit), at Month 6, Month 12, and Month 18 follow-ups.
  Minimum: 45, maximum: 315, a higher score means a better outcome.
Number of incidental diagnoses of Mild Cognitive Impairment (MCI) and dementia, according to National Institute on Aging-Alzheimer's Association (NIA-AA) criteria | Through study completion, an average of 2 years.
  A higher number means a worse outcome.
Composite score of processing speed and attention | The score will be taken at Baseline visit (Day 0 of second phase, which should be indicatively within 30 days of Screening visit), at Month 6, Month 12, and Month 18 follow-ups.
  z-score without a maximum or minimum value, a higher z-score means a better outcome.
Composite score of executive functions | The score will be taken at Baseline visit (Day 0 of second phase, which should be indicatively within 30 days of Screening visit), at Month 6, Month 12, and Month 18 follow-ups.
  z-score without a maximum or minimum value, a higher z-score means a better outcome.
Composite memory score | The score will be taken at Baseline visit (Day 0 of second phase, which should be indicatively within 30 days of Screening visit), at Month 6, Month 12, and Month 18 follow-ups.
  z-score without a maximum or minimum value, a higher z-score means a better outcome.
Composite language score | The score will be taken at Baseline visit (Day 0 of second phase, which should be indicatively within 30 days of Screening visit), at Month 6, Month 12, and Month 18 follow-ups.
  z-score without a maximum or minimum value, a higher z-score means a better outcome.
Composite score of general cognitive assessment | The score will be taken at Baseline visit (Day 0 of second phase, which should be indicatively within 30 days of Screening visit), at Month 6, Month 12, and Month 18 follow-ups.
  z-score without a maximum or minimum value, a higher z-score means a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS San Gerardo dei Tintori, Monza, Italy

REFERENCES:
- [Derived] Sala G, Cuffaro L, Pozzi FE, Andreoni S, Bazzini C, Conti E, Zoia CP, Beretta S, Tremolizzo L, Bellelli G, Okoye C, Ferrara MC, De Luca A, Lenti R, Mantuano P, Pontrelli P, Stasi A, Defazio G, Solfrizzi V, Crudele L, Airoldi C, Chiaradonna F, Longhese MP, Messina G, Natalello A, Orlandi I, Aloisi A, Capone S, Ingannato A, Nacmias B, Capello D, Mangialasche F, Ferrarese C. Multi-pathway blood biomarkers to target and monitor multidimensional prevention of cognitive and functional decline (nested in the IN-TeMPO study framed within the world-wide FINGERS network). Front Aging Neurosci. 2025 May 7;17:1581892. doi: 10.3389/fnagi.2025.1581892. eCollection 2025. PMID 40400914